CLINICAL TRIAL: NCT03598816
Title: A Randomized Phase II PIVOT-RCC (PolyImmune {Durvalumab (MEDI4736) and Tremelimumab} & Vaccine Orchestrated Treatment for Patients With Advanced/Metastatic Renal Cell Carcinoma) Trial
Brief Title: PolyImmune {Durvalumab (MEDI4736) and Tremelimumab} & Vaccine Orchestrated Treatment for Patients With Advanced/Metastatic Renal Cell Carcinoma
Acronym: PIVOT-RCC
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: FDA Contingencies unresolved
Sponsor: Washington University School of Medicine (Other)
Collaborators: MedImmune LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 202003083
Record Dates: First submitted 2018-07-16; First posted 2018-07-26 (Actual); Last update posted 2020-08-13 (Actual); Status verified 2020-08

CONDITIONS: Renal Cell Carcinoma
MeSH Terms: conditions — Carcinoma, Renal Cell | interventions — durvalumab; tremelimumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Arm 1: Durvalumab + Tremelimumab + Neoantigen DNA Vaccine (Experimental): * All patients will receive durvalumab intravenous (IV) at a dose of 10 mg/kg over the course of 60 minutes given every 2 weeks (on Days 1 and 15 of each 28-day cycle) for a total of 8 doses. Durvalumab will be given thereafter as monotherapy at a dose of 209 mg/kg over the course of 60 minutes given every 4 weeks (on Day 1 of each 28-day cycle) for a total of 4 doses
  * All patients will receive tremelimumab at a dose of 1 mg/kg over the course of 60 minutes given every 4 weeks (on Day 1 of each 28-day cycle) for a total of 4 cycles
  * The first vaccination will take place two weeks after confirmed disease progression on targeted therapy. This will be Day 1 of the first 28-day cycle of treatment with durvalumab and tremelimumab
  * The schedule of vaccination is Cycle 1 Day 1, Cycle 1 Day 15, Cycle 2 Day 1, Cycle 3 Day 1, Cycle 4 Day 1, and Cycle 5 Day 1 (for a total of 6 doses)
  Interventions: Drug: Durvalumab; Drug: Tremelimumab; Device: TDS-IM v1.0 System; Biological: Neoantigen DNA Vaccine; Procedure: Research blood draw
- Arm 2: Durvalumab + Tremelimumab (Experimental): * All patients will receive durvalumab IV at a dose of 10 mg/kg over the course of 60 minutes given every 2 weeks (on Days 1 and 15 of each 28-day cycle) for a total of 8 doses. Durvalumab will be given thereafter as monotherapy at a dose of 209 mg/kg over the course of 60 minutes given every 4 weeks (on Day 1 of each 28-day cycle) for a total of 4 doses
  * All patients will receive tremelimumab at a dose of 1 mg/kg over the course of 60 minutes given every 4 weeks (on Day 1 of each 28-day cycle) for a total of 4 cycles.
  Interventions: Drug: Durvalumab; Drug: Tremelimumab; Procedure: Research blood draw

INTERVENTIONS:
Drug: Durvalumab — -Durvalumab infusion will start approximately 1 hour (maximum 2 hours) after the end of the tremelimumab infusion
  Other Names: Imfinzi; MEDI4736
Drug: Tremelimumab — -Tremelimumab will be administered first
Device: TDS-IM v1.0 System — -Integrated electroporation device
  Arms: Arm 1: Durvalumab + Tremelimumab + Neoantigen DNA Vaccine
Biological: Neoantigen DNA Vaccine — -At each vaccination time point, patients will receive two injections of the neoantigen DNA vaccine, one injection into each deltoid or lateralis.
  Arms: Arm 1: Durvalumab + Tremelimumab + Neoantigen DNA Vaccine
Procedure: Research blood draw — -Baseline, C2D1, C3D1, C5D1, C7D1, and C9D1

SUMMARY:
Reported in the 2018 NEJM (378; 1277) article, the combination of checkpoint inhibitors ipilimumab (anti-CTLA-4 antibody) and nivolumab (anti-PD-1 antibody) phase III trial Checkmate 214 demonstrated statistically significant (P<0.0001) improvement of overall response rate (ORR) at 42% (95% confidence interval (CI), 37-47%) compared to standard of care (SOC) sunitinib at 27% (95% CI, 22-31%) in treatment naïve advanced or metastatic clear cell renal cell carcinoma (ccRCC). This study also showed increased survival benefit of Ipi+Nivo over sunitinib in the IMDC intermediate-poor risk ccRCC patients. Accordingly, the Ipi+Nivo was just approved by U.S. FDA in April 2018 for treating metastatic ccRCC. Hence, the investigators hypothesized that the combination of durvalumab and tremelimumab is similarly efficacious in advanced or metastatic RCC. Furthermore, the investigators also hypothesize that the administration of personalized neoantigen DNA vaccine will further enhance anti-tumor immune response in RCC.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of histologically confirmed metastatic/advanced (inoperable) renal cell carcinoma with clear cell or non-clear cell histology.
* Measurable disease by RECIST 1.1
* Must have progressed on at least one but no more than two lines of targeted therapies or have increasing incidences and intolerability of ≥ Gr.2 AE (CTCAE) toxicity from ongoing targeted therapies. Targeted therapies that cause immediate toxicities and result in discontinuation of treatment within 4 weeks after the start of individual treatments are not considered as progression.
* Consented for genome sequencing and data sharing.
* Life expectancy of at least 12 weeks.
* At least 18 years of age.
* Karnofsky performance status ≥ 70%
* Normal bone marrow and organ function as defined below:

  * Absolute neutrophil count ≥ 1,000/mcL
  * Platelets ≥ 75,000/mcL
  * Hemoglobin ≥ 9.0 g/dL
  * Serum bilirubin ≤ 1.5 x institutional upper limit of normal (IULN). This does not apply to patients with confirmed Gilbert's syndrome, who will be allowed in consultation with their physician
  * AST(SGOT)/ALT(SGPT) ≤ 2.5 x IULN; for patients with hepatic metastases, ALT and AST ≤ 4 x IULN
  * Measured creatinine clearance > 40 mL/min or calculated creatinine clearance > 40 mL/min as determined by Cockcroft-Gault using actual body weight
* Evidence of post-menopausal status or negative urinary or serum pregnancy test for female pre-menopausal patients. Women will be considered post-menopausal if they have been amenorrheic for 12 months without an alternative medical cause. The following age-specific requirements apply:

  * Women <50 years of age would be considered post-menopausal if they have been amenorrheic for 12 months or more following cessation of exogenous hormonal treatments and if they have luteinizing hormone and follicle-stimulating hormone levels in the post-menopausal range for the institution or underwent surgical sterilization (bilateral oophorectomy or hysterectomy).
  * Women ≥50 years of age would be considered post-menopausal if they have been amenorrheic for 12 months or more following cessation of all exogenous hormonal treatments, had radiation-induced menopause with last menses >1 year ago, had chemotherapy-induced menopause with last menses >1 year ago, or underwent surgical sterilization (bilateral oophorectomy, bilateral salpingectomy or hysterectomy).
* Ability to understand and willingness to sign an IRB approved written informed consent document (or that of legally authorized representative, if applicable).

Exclusion Criteria:

* Received any immuno-oncology agents including, but not limited to, other anti CTLA-4, including tremelimumab anti-PD-1, anti-PD-L1 including durvalumab, and anti-programmed cell death ligand 2 (anti-PD-L2) antibodies, excluding therapeutic anticancer vaccines. Patients with prior adjuvant or neoadjuvant treatment of targeted therapies for RCC are eligible.
* A history of other malignancy ≤ 2 years previous with the exception of basal cell or squamous cell carcinoma of the skin which were treated with local resection only or carcinoma in situ of the cervix.
* Currently receiving any other investigational agents.
* Spinal cord compression or clinically active central nervous system metastasis, defined as untreated and symptomatic, or requiring therapy with corticosteroids. Subjects with treated brain metastasis that are no longer symptomatic may be included. A minimum of 2 weeks must have elapsed between the end of radiation and the study enrollment.
* A history of allergic reactions attributed to compounds of similar chemical or biologic composition to durvalumab, tremelimumab, vaccines, or other agents used in the study.
* Receipt of live attenuated vaccine within 30 days prior to the first dose of study treatment.
* Any unresolved toxicity NCI CTCAE Grade ≥2 from previous anticancer therapy with the exception of alopecia, vitiligo, and the laboratory values defined in the inclusion criteria -Patients with Grade ≥2 neuropathy will be evaluated on a case-by-case basis after consultation with the Study Physician.
* Patients with irreversible toxicity not reasonably expected to be exacerbated by treatment with durvalumab or tremelimumab may be included only after consultation with the Study Physician.
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, uncontrolled hypertension, unstable angina pectoris, cardiac arrhythmia, interstitial lung disease, or serious chronic gastrointestinal conditions associated with diarrhea.
* Mean QT interval corrected for heart rate using Fridericia's formula (QTcF) ≥470 ms calculated from 3 ECGs (within 15 minutes at 5 minutes apart).
* History of leptomeningeal carcinomatosis.
* History of syncopal or vasovagal episode as determined by medial record and history in the 6-month period prior to first vaccination administration.
* Individuals in whom a skinfold measurement of the cutaneous and subcutaneous tissue for eligible injection sites (left and right medial deltoid region) exceeds 40 mm.
* Individuals in whom the ability to observe possible local reactions at the eligible injection sites (deltoid region) is, in the opinion of the investigator, unacceptably obscured due to a physical condition or permanent body art.
* Therapeutic or traumatic metal implant in the skin or muscle of either deltoid region.
* Any current chronic or active neurologic disorder, including seizures and epilepsy, requires active medical management.
* Current use of any electronic stimulation device, such as cardiac demand pacemakers, automatic implantable cardiac defibrillator, nerve stimulators, or deep brain stimulators.
* Major surgical procedure (as defined by the PI) within 28 days prior to the first dose of durvalumab and tremelimumab. Note: Local surgery of isolated lesions for palliative intent is acceptable.
* History of allogenic organ transplantation.
* Active or prior documented autoimmune or inflammatory disorders (including inflammatory bowel disease [eg, colitis or Crohn's disease], diverticulitis [with the exception of diverticulosis], systemic lupus erythematosus, Sarcoidosis syndrome, or Wegener syndrome [granulomatosis with polyangiitis, Graves' disease, rheumatoid arthritis, hypophysitis, uveitis, etc]). The following are exceptions to this criterion:

  * Patients with vitiligo or alopecia
  * Patients with hypothyroidism (eg, following Hashimoto syndrome) stable on hormone replacement
  * Any chronic skin condition that does not require systemic therapy
  * Patients without active disease in the last 5 years may be included but only after consultation with the study physician
  * Patients with celiac disease controlled by diet alone
* History of active primary immunodeficiency
* Active infection including tuberculosis (clinical evaluation that includes clinical history, physical examination and radiographic findings, and tuberculosis testing in line with local practice), hepatitis B (known positive HBV surface antigen (HBsAg) result), hepatitis C, or human immunodeficiency virus (positive HIV 1/2 antibodies). Patients with a past or resolved HBV infection (defined as the presence of hepatitis B core antibody [anti-HBc] and absence of HBsAg) are eligible. Patients positive for hepatitis C (HCV) antibody are eligible only if polymerase chain reaction is negative for HCV RNA.
* Current or prior use of immunosuppressive medication within 14 days before the first dose of durvalumab or tremelimumab. The following are exceptions to this criterion:

  * Intranasal, inhaled, topical steroids, or local steroid injections (eg, intra articular injection)
  * Systemic corticosteroids at physiologic doses not to exceed 10 mg/day of prednisone or its equivalent
  * Steroids as premedication for hypersensitivity reactions (eg, CT scan premedication)
* Pregnant and/or breastfeeding. Women of childbearing potential must have a negative serum/urine pregnancy test within 14 days of study entry. All patients must be willing to employ effective birth control from screening to 90 days after the last dose of durvalumab monotherapy or 180 days after the last dose of durvalumab + tremelimumab combination therapy.
* Known HIV-positive status. These patients are ineligible because of the potential inability to generate an immune response to vaccines.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-08-31 (Estimated); Primary Completion 2022-12-31 (Estimated); Study Completion 2024-05-31 (Estimated)

PRIMARY OUTCOMES:
Safety of the combination of durvalumab & tremelimumab with or without neoantigen DNA vaccine when given to patients with renal cell carcinoma as measured by the percentage of patients with adverse events of grade 3 or higher | Completion of cycle 1 (4 weeks)
  * As graded by the revised NCI Common Terminology Criteria for Adverse Events (CTCAE) version 5.0
  * Only adverse events that are possibly, likely, or probably related to the drug or drug combinations

SECONDARY OUTCOMES:
Response rate in patients with renal cell carcinoma treated with durvalumab and tremelimumab with or without neoantigen DNA vaccine by RECIST 1.1 as measured by percentage of patients with radiographic complete response or partial response | Through completion of treatment (estimated to be 32-36 weeks)
  * Complete response: Disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm. Disappearance of all non-target lesions and normalization of tumor marker level.
  * Partial response: At least a 30% decrease in the sum of the diameters of target lesions, taking as reference the baseline sum diameters
Rate of progression-free survival (PFS) in patients with renal cell carcinoma treated with durvalumab and tremelimumab with or without neoantigen DNA vaccine | Through 6 months after completion of treatment (estimated to be 15 months)
  * PFS defined as from time of randomization to time of progression or death due to any cause, whichever earlier and if no progression or death, to time of last follow up
  * Progressive disease: At least a 20% increase in the sum of the diameters of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study). In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm. (Note: the appearance of one or more new lesions is also considered progressions).
Rate of overall survival (OS) in patients with renal cell carcinoma treated with durvalumab and tremelimumab with or without neoantigen DNA vaccine | Through 6 months after completion of treatment (estimated to be 15 months)
  -OS) defined as from time of randomization to time of death due to any cause and if patients are still alive at end of the study, to the time of last follow up

CONTACTS AND LOCATIONS:
Overall Officials: James J Hsieh, M.D., Ph.D., Principal Investigator — Washington University School of Medicine

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://www.siteman.wustl.edu